CLINICAL TRIAL: NCT02061449
Title: A Pilot Study of a Novel Multimodality Immuno-Chemotherapy Platform for Patients With Advanced Cutaneous T Cell Lymphoma
Brief Title: Poly ICLC, Radiation, and Romidepsin for Advanced Cutaneous T Cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: NYU Langone Health (Other)
Collaborators: Ludwig Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-00686
Record Dates: First submitted 2014-02-11; First posted 2014-02-12 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Cutaneous T-cell Lymphoma
Keywords: Toll-like receptor agonist; immunostimulation
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — romidepsin; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Initiating therapy with Romidepsin (Arm A) (Experimental): Patients who are starting therapy with Romidepsin (intravenously on days 1, 8, and 15 of every 21-day cycle or alternate schedule per treating physician) also receive focal lesional radiation on days 1,3, and 5 without (level 1) or with (level 2) Poly ICLC (subcutaneously on days 1, 3, and 5) on the first cycle.
  Interventions: Drug: Romidepsin; Drug: Poly ICLC; Radiation: Focal lesional radiation
- treatment with Romidepsin with SD or PR (Arm B) (Experimental): Patients with stable disease on the treatment with Romidepsin (intravenously on days 1, 8, and 15 of every 21-day cycle or alternate schedule per treating physician) also receive focal lesional radiation on days 1,3, and 5 without (level 1) or with (level 2) Poly ICLC (subcutaneously on days 1, 3, and 5) on the first cycle.
  Interventions: Drug: Romidepsin; Drug: Poly ICLC; Radiation: Focal lesional radiation

INTERVENTIONS:
Drug: Romidepsin
  Other Names: Istodax; FK228; FR901228
Drug: Poly ICLC
Radiation: Focal lesional radiation

SUMMARY:
This study evaluates the safety and tolerability of the addition of immunostimulatory therapy consisting of focal radiation with or without the Toll-like receptor (TLR) agonist Poly ICLC in patients with cutaneous T-cell lymphoma (CTCL) receiving concurrent therapy with the histone deacetylase inhibitor (HDACI) Romidepsin.

DETAILED DESCRIPTION:
Histone deacetylase inhibitors in epigenetic therapy are one of the most active anti-tumor agents in patients with relapsed and refractory CTCL despite their suppressive effects on T cell function, yet the overall response rate and response duration with these agents remains suboptimal. Immune stimulatory agents may be the ideal therapy to combine with HDACI. To date, no one has evaluated whether the abscopal effect of radiation with and without the additional immune stimulation of a TLR-3 agonist can augmented the efficacy of anti-tumor directed epigenetic therapy in mycosis fungoides (MF) patients. The investigators hypothesize that a combined modality immuno-chemotherapy may be highly effective in patients with advanced MF.

This is a phase I study. It involves two arms of patients (A and B) who will be treated following a standard 3+ 3 design. Patients on Arm A are the ones who are initiating HDACI therapy, and patients on Arm B are the ones with stable disease or partial response with HDACI treatment. Both groups receive HDACI, plus at level 1, focal lesional radiation; at level 2, radiation in combination with Poly ICLC. Each arm will be evaluated and escalated independently.

ELIGIBILITY:
Inclusion Criteria:

* Must have prior biopsy at any time point diagnostic for confirmed MF stage IIA-IVA, and must have failed at least one standard therapy (topical or systemic).
* Must have a skin lesion of at minimum 2 cm, in a location amenable to radiation and a minimum of 2 additional measurable skin lesions distant from the radiation site.
* Must be either initiating therapy with romidepsin (Arm A) or currently receiving romidepsin with documented stable disease (SD) or partial response (PR) (Arm B).
* Patient may have had any prior topical or systemic therapy except for total electron beam irradiation. Patients must be a minimum of 2 weeks from topical therapy and 4 weeks from systemic therapies, phototherapy, or local radiation therapy before enrollment except for HDACI if they are in Arm B. Patients are allowed to take weak potency topical corticosteroids if patient has been on a stable dose for more than a month.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >70%)
* Life expectancy of greater than 6 months
* Patients must have normal organ and marrow function as defined below:

  * leukocytes >=2,500/mcL
  * absolute neutrophil count >=1,000/mcL
  * platelets >=50,000/mcL
  * total bilirubin: within normal institutional limits
  * AST(SGOT, aspartate aminotransferase)/ALT(SGPT, alanine aminotransferase) =<2.5 X institutional upper limit of normal
  * creatinine: within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
* Age >=18 years
* The effects of focal radiation and HDACI on the developing human fetus are unknown. For this reason and because agents as well as other therapeutic agents used in this trial are known to be tetragenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks, or topical therapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Patients are allowed to take weak potency topical corticosteroids if patient has been on a stable dose for more than a month.
* Patients who are receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to HDACI, TLR-agonist, or patients with known history of pre-existing auto-immune disease.
* Concurrent therapy with systemic corticosteroids or other immunosuppressive medications.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study HDACI is a class agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with HDACI, breastfeeding should be discontinued if the mother is treated with HDACI and radiation. Woman of childbearing age and men sexually active with woman of childbearing age must agree to an acceptable method of birth control (double barrier) while on study.
* Patients with known HIV infection are ineligible because this immunomodulatory therapy requires a normal and functional T cell repertoire. If this study is found to be safe, effective, and immunogenic, HIV positive patients may be included in future studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 21 days
  Adverse events and dose-limiting toxicities will be graded using National Cancer Institute's Common Toxicity Criteria for Adverse Effects (CTCAE) 4.0.

SECONDARY OUTCOMES:
Overall response rate | Up to 12 months
  Defined as the percentage of patients who achieve complete response or partial response. The response is evaluated based on Modified Severity weighted Assessment Tool (MSWAT) criteria.
Median progression-free survival | up to 12 months
  Progression-free survival is defined as the time from study entry to the first documented of tumor progression ot death due to any cause whichever comes first.
Median overall survival | up to 12 months
  Overall survival is described as the time from study entry to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Diefenbach, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Cancer Institute, New York, New York, United States